CLINICAL TRIAL: NCT01288599
Title: Single Port Laparoscopy Versus Conventional Laparoscopy for Benign Adnexal Disease - A Randomized Controlled Trial.
Brief Title: Single Versus Conventional Laparoscopy for Benign Adnexal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Laparoscopy SSK
Record Dates: First submitted 2010-11-18; First posted 2011-02-02 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2011-02

CONDITIONS: Ovarian Cyst
Keywords: Laparoscopy; Randomized; Single port access; Adnexal disease; LESS
MeSH Terms: conditions — Ovarian Cysts; Adnexal Diseases | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single port access laparoscopy (Experimental): Single port access laparoscopy for benign adnexal disease.
  Interventions: Procedure: Laparoscopic surgery
- Conventional laparoscopy (Active Comparator): Conventional laparoscopy for benign adnexal disease.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — Laparoscopic surgery where adnexectomy or cystectomy is performed.

SUMMARY:
Keyhole surgery for adnexal disease has traditionally been performed using three or four small incisions. The last years a new operating method has been introduced. This method makes use of only one incision of 2 cm in the umbilicus. This method is less invasive, and it might benefit the patient through less postoperative pain and a higher satisfaction with the cosmetic result. So far, many studies have shown that this new method is feasible for adnexal disease, but its superiority compared to conventional laparoscopy is to be proven. This study aims to show this difference.

The investigators aim to compare experienced postoperative pain and use of analgesics in patients undergoing single port laparoscopy for benign adnexal disease with conventional laparoscopy. The investigators hypothesize that the patients will experience less postoperative pain and use less analgesic in the single port laparoscopy group.

Further, the investigators aim to compare the satisfaction with the cosmetic results in the two groups. In addition, blood loss, operating time, complications and conversion to conventional laparoscopy will be registered in the two groups.

DETAILED DESCRIPTION:
Although there are many reports indicating that single port laparoscopy for benign adnexal disease is feasible, there have to date not been published any randomized studies proving a superior outcome compared to conventional laparoscopy.

Theoretically, there are several advantages with a single port access. Because only one incision is made in place of several, less postoperative pain could be expected. The incision made is slightly larger (2 cm) than the ones used in conventional laparoscopy. It could therefore be easier to evacuate carbon dioxide gas (CO2) out of the abdomen after the operation, resulting in less shoulder tip pain, which is a common discomfort postoperatively. Carbon dioxide gas is considered to be responsible for postoperative shoulder tip pain due to peritoneal stretching and diaphragmatic irritation (Alexander et al. 1987, Sarli et al. 2000). The better cosmetic result due to only one incision is apparent. If this improvement makes a different for the patients, is yet to be proven.

There might be fewer complications with single-port laparoscopy compared to conventional laparoscopy. As mentioned above, serious complications like bowel and vessel injury, mostly occurring when Verres needle or a trocar is introduced through the abdominal wall. By reducing the number of trocars introduced, these complications might occur less commonly.

Performing a randomized controlled trial will bring more knowledge to whether single port laparoscopy for benign adnexal disease will truly benefit the patients compared to the established operating method for this condition.

Surgical technique:

Preoperatively, all patients will be given paracetamol 1.5 grams, diclofenac 100 mg and oxycodone 10 mg as a single dose orally analgesics. Under general anaesthesia and endotracheal intubation the patient will be positioned in the dorsal lithotomy position with both legs supported in Allen stirrups and their arms resting alongside the body. An orogastric tube will be placed to decompress the stomach and a Foley catheter will be placed in the bladder.

In the single port laparoscopy group, 10 ml of 0.5 % bupivacaine hydrochloride (Marcain®) will be injected subcutaneously as local anaesthetic before a 2 cm vertical incision (measured with a sterile ruler) will be made through the umbilicus. The rectus fascia will be sharply incised and a single multiport trocar (Laparo-Endoscopic Single-Site Surgery, Olympus Winter & IBE GMBH, Hamburg, Germany) will be introduced via an introducer device in the peritoneal cavity. This port has an insufflation channel that allows carbon dioxide insufflation with the pressure set at 12 mm Hg. To obtain intrabdominal visualization, a 5-mm 30º telescope (EndoEye, Olympus Winter & IBE GMBH, Hamburg, Germany) will be used. A diagnostic peritoneal lavage will be performed. The patient will be placed in a Trendelenburg position. Curved hand instruments (HiQ LS, Olympus Winter & IBE GMBH, Hamburg, Germany) will be used to provide efficient retraction to optimize surgical exposure. A straight bipolar diathermy and scissors will be used to extirpate the cyst or remove the adnexa. After cystectomy or adnexectomy has been performed, the excised tissue will be removed through the multichannel port. Larger masses will be placed in 10-mm Endo Catch™ Gold (Covidien, Norwalk Connecticut, USA) to avoid spillage. If necessary, decompression of pelvic masses will be done with a 14-gauge angiocath needle at the umbilical incision after removal of the single port device. After removal of the tissue the multichannel access port will be opened to evacuate CO2. The port will be removed and the fascia will be sutured with Polysorb 0 suture. The skin will be closed using abrupt intracutaneous Polysorb 3-0 sutures.

In the conventional laparoscopy group, 5 ml of 0.5 % bupivacaine hydrochloride (Marcain®) will be injected as local anaesthetic before a 1 cm incision will be made in the umbilicus. Abdominal access will be gained by using an open entry technique. A suture will be placed in the fascia with Polysorb 0. Carbon dioxide will be insufflated through this port with a pressure set at 12 mm Hg. 5 ml of 0.5 % bupivacaine hydrochloride (Marcain®) will be injected at each of the places for three additional ports. Two 5-mm accessory Versaport™ Blade less trocars (Covidien, Norwalk Connecticut, USA) will be inserted in the lower right and left quadrant and a 12-mm Versaport™ Blade less trocar will be inserted in the midline, approximately 2 cm above the symphysis. Diagnostic peritoneal lavage will be performed. Cystectomy or adnexectomy will be performed using bipolar diathermy, scissors and a grasper. The tissue will be placed in 10-mm Endo Catch™ Gold (Covidien, Norwalk Connecticut, USA) and removed through the incision in the midline above the symphysis. If necessary, decompression of pelvic masses will be done with a 14-gauge angiocath needle and the skin incision would be extended to a maximum of 2 cm. The fascia in the midline incision above the symphysis will be sutured with Polysorb 0 using the Endoclose® hook (Covidien, Norwalk Connecticut, USA). The fascia in the umbilicus will be closed with the earlier placed suture and the skin in the midline incisions will be closed using abrupt intracutaneous Polysorb 3-0 sutures. The incisions in the right en left fossa will be closed using Steristrips™.

After the operation, the patients will receive analgesics on request. Their pain scores will be registered on a linear 10 cm visual analogue scale at 6 hours and 24 hours after the operation. They will also be asked if they experience shoulder tip pain. This pain will be registered after 6 hours and 24 hours. The use of analgesics while admitted at the hospital will be registered. They will be discharged from the hospital the first postoperative day. The patients will be contacted and asked about their use of analgesics for the next two days.

Two months after the operation, the patients will be asked to rate their satisfaction with the cosmetic result on a five point scale ranging from extremely unsatisfied to extremely satisfied. There will also be taken a picture of the scar in the umbilicus, which will be rated according to the Manchester scar scale (Beausang et al. 1998).

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years.
* ASA score 1 or 2.
* Presumed benign ovarian disease or a hereditary cancer risk.
* Ovarian cyst ≤ 6 cm.

Exclusion Criteria:

* Ovarian cyst > 6 cm.
* Endometrioma.
* Endometriosis.
* History of chronic pelvic pain.
* Known severe intra abdominal adhesions.
* Daily use of analgesics.
* Inability to understand Norwegian or English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 hours
  Experienced pain over the last six hours measured on a VAS scale.

SECONDARY OUTCOMES:
Satisfaction with cosmetic result | 2 months postoperatively
  Satisfaction with cosmetic result, self reported and based on the Manchester scar scale.
Operation time | 0 hours after the operation
  Operating time in minutes.
Blood loss | 0 hours after the operation
  Estimated blood loss in ml.
Complications | Two months
  Complications during surgery and late complications.
Shoulder tip pain | 24 hours
  Experienced shoulder tip pain over the last 24 hours measured on a VAS scale.
Postoperative pain | 24 hours
  Experienced pain over the last 24 hours measured on a VAS scale.

CONTACTS AND LOCATIONS:
Locations (1):
- SorlandetHF Hospital, Kristiansand, Norway

REFERENCES:
- [Derived] Hoyer-Sorensen C, Vistad I, Ballard K. Is single-port laparoscopy for benign adnexal disease less painful than conventional laparoscopy? A single-center randomized controlled trial. Fertil Steril. 2012 Oct;98(4):973-9. doi: 10.1016/j.fertnstert.2012.06.016. Epub 2012 Jul 4. PMID 22769732